CLINICAL TRIAL: NCT06406803
Title: The Impact of Physical Activity Versus Dietary Energy Restriction on Prostate Tumour and Muscle Tissue Protein Synthesis in Vivo in Prostate Cancer Patients
Brief Title: The Impact of Physical Activity Versus Dietary Energy Restriction on Tumour and Muscle Protein Synthesis in Prostate Cancer Patients
Acronym: DIRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: f/2023/047
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary energy restriction (Experimental)
  Interventions: Behavioral: Dietary energy restriction
- Daily exercise (Experimental)
  Interventions: Behavioral: Daily exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Dietary energy restriction — Patients enrolled in the dietary energy restriction group will reach an energy deficit of 40% only through reduced dietary intake.
  Arms: Dietary energy restriction
Behavioral: Daily exercise — Patients in the daily exercise group will reach an energy deficit of 40% through reduced dietary intake and increased physical activity (exercise).
  Arms: Daily exercise

SUMMARY:
Background: Prostate cancer is the second most common cancer and the fifth leading cause of death in men worldwide. Tumour growth is attributed to disproportionately greater protein synthesis rates relative to protein breakdown rates. Tumour protein synthesis is modulated by several factors, including energy availability, blood flow, and hormone concentrations (e.g., IGF-1). Lifestyle modifications are rapidly becoming recognized as important adjunct therapeutic approaches to slow cancer development and enhance treatment efficacy. Dietary energy restriction is a 30-50% reduction in food intake, which induces an energy deficit and has been shown to attenuate tumour growth in rodent models. Muscle mass often declines during cancer treatment and negatively impacts treatment success rates and recovery. One drawback to dietary energy restriction is that it may accelerate declines in skeletal muscle mass and strength in cancer patients. Exercise also induces an energy deficit by increasing energy expenditure. In addition, exercise alters blood flow and releases circulating molecules, which appear to lower tumour protein synthesis rates. Exercise increases muscle protein synthesis rates, which would provide further benefits to cancer patients by helping to maintain skeletal muscle mass. Despite their promising therapeutic properties, the clinical efficacy of dietary energy restriction and exercise has not been directly determined in vivo in cancer patients.

Hypothesis and Objectives: The objective of this study is to compare the impact of dietary energy restriction versus (isocaloric) daily exercise on muscle, prostate, and prostate tumour protein synthesis rates over a 7-day period in vivo in prostate cancer patients.

It is hypothesized that 1) dietary energy restriction will lower both prostate tumour and muscle tissue protein synthesis rates and that 2) daily exercise will lower prostate tumour protein synthesis rates but increase muscle protein synthesis rates in prostate cancer patients.

Setting and Methods: Forty-five prostate cancer patients scheduled to undergo radical prostatectomy will be randomly assigned to one of three groups. The first group will undergo 7 days of dietary energy restriction (40% less food intake). The second group will perform 7 days of daily exercise and mild dietary energy restriction resulting in a total energy deficit of 40%. The third group will follow their regular diet and physical activity (control group). The research team will provide all aspects of the intervention (standardized meals, personalized exercise supervision). Patients will ingest deuterium-labelled water (2H2O) throughout the intervention period. After 7 days, patients will undergo a radical prostatectomy, during which tumour tissue, skeletal muscle tissue, and blood will be collected. Deuterium (2H-alanine) incorporation into the tissue samples will be measured to assess prostate tumour and skeletal muscle tissue protein synthesis rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer (Stages I-III)
* Scheduled to undergo a prostatectomy
* BMI between 18.5-35 kg/m2

Exclusion Criteria:

* Receiving pre-operative chemo, hormonal, radio therapy
* Physically unable to perform the exercise program
* Performing >300 min of moderate-vigorous physical activity per week (e.g., running, road cycling, swimming).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Tumour protein synthesis rates | 7 days pre-operatively
  Measured using the deuterated water (2H2O) method
Muscle protein synthesis rates | 7 days pre-operatively
  Measured using the deuterated water (2H2O) method

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium